CLINICAL TRIAL: NCT00248495
Title: Molecular and Genetic Changes in Patients With Resectable Non-Small Cell Lung Cancer (NSCLC) Following Neoadjuvant Chemotherapy With Cisplatin and Alimta - Phase II Study
Brief Title: Pemetrexed Disodium and Cisplatin in Treating Patients Who Are Undergoing Surgery for Stage I, Stage II, or Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000441025; RPCI I-31104; NCT01731626 (obsolete NCT alias)
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage II non-small cell lung cancer; stage I non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Pemetrexed; Chemotherapy, Adjuvant; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neoadjuvant chemotherapy (Experimental): Patients receive pemetrexed disodium IV over 10 minutes followed by cisplatin IV over approximately 1 hour on day 1. Treatment repeats every 21 days for 3 courses
  Interventions: Drug: cisplatin; Drug: pemetrexed disodium; Procedure: adjuvant therapy; Procedure: conventional surgery; Procedure: neoadjuvant therapy

INTERVENTIONS:
Drug: cisplatin — Given IV
Drug: pemetrexed disodium — Given IV
Procedure: adjuvant therapy — Metastasis prevention/control
Procedure: conventional surgery — Undergoing tissue removal
Procedure: neoadjuvant therapy — Tumor Reduction

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as pemetrexed disodium and cisplatin work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) and giving them before and after surgery may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving pemetrexed disodium and cisplatin before and after surgery works in treating patients with stage I, stage II, or stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the pathologic complete response in patients with stage IB-IIIB non-small cell lung cancer treated with neoadjuvant chemotherapy comprising pemetrexed disodium and cisplatin followed by surgery and adjuvant pemetrexed disodium and cisplatin.

Secondary

* Determine the adverse events of this regimen in these patients.
* Determine the overall and disease-free survival of patients treated with this regimen.
* Correlate response with the presence or absence of ERCC1 and DHFR, thymidylate synthase, DPD, and GARFT in patients treated with this regimen.
* Correlate the fragile site on chromosome 12 within the SMRT gene with metastasis after definitive treatment with this regimen in these patients.

OUTLINE:

* Neoadjuvant chemotherapy: Patients receive pemetrexed disodium IV over 10 minutes followed by cisplatin IV over approximately 1 hour on day 1. Treatment repeats every 21 days for 3 courses. Patients are then evaluated for disease resectability. Patients with no evidence of disease progression proceed to thoracotomy within the next 28-48 days.
* Thoracotomy: Patients found to have unresectable disease during thoracotomy receive further treatment off study. Patients with resectable disease undergo complete surgical resection of the tumor. Forty to eighty days later, patients proceed to adjuvant chemotherapy.
* Adjuvant chemotherapy: Patients receive pemetrexed disodium and cisplatin as before for 2 courses.

Patients with progressive disease after completion of neoadjuvant chemotherapy are followed every 6 months. All other patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 38 patients will be accrued for this study over 6.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Microscopically confirmed non-small cell lung cancer

  * Stage IB (T2, N0, M0), IIA (T1, N1, M0), IIB (T2, N1, M0 or T3, N0, M0), or IIIA (T1-3, N1-2, M0) disease
  * Satellite lesions in one lobe (T4) (stage IIIB) allowed
* Meets 1 of the following criteria:

  * Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 10 mm in the longest diameter
  * Evaluable disease, defined as lesions on chest CT scan that are not measurable (e.g., ill-defined masses or mediastinal or hilar adenopathy)
* No metastatic disease except peribronchial/hilar lymph nodes (N1) or ipsilateral/subcarinal mediastinal lymph nodes (N2)

  * No N3 lymph nodes (e.g., contralateral mediastinal/hilar or supraclavicular/scalene) by CT scan or positron emission tomography (PET) scan AND mediastinoscopy
  * No T4 primary tumor (e.g., mediastinal invasion)
* No malignant pleural effusion

  * Nonmalignant effusions (i.e., negative cytology, non-bloody, and transudate) allowed
  * Effusions visible only by CT scan and not large enough for safe thoracentesis allowed
* No exudative effusion, defined by 1 of the following criteria:

  * Pleural fluid protein:serum protein ratio > 0.5
  * Pleural fluid lactic dehydrogenase (LDH):serum LDH ratio ≥ 0.6
  * Pleural fluid LDH > 200 IU/L
* No more than 1 area of fludeoxyglucose (FDG) uptake outside the area of the primary lung tumor OR evidence of malignant pleural disease as evidenced by pleural nodules by PET scan

  * Single areas of FDG uptake will be further evaluated (e.g., by biopsy) for metastatic disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* SGOT or SGPT ≤ 1.5 times upper limit of normal

Renal

* Creatinine clearance ≥ 45 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No other active malignancy within the past 2 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No psychological, familial, sociological, or geographical situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for lung cancer

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for lung cancer

Surgery

* No prior surgery for lung cancer
* At least 12 weeks since prior major surgery to the chest and abdomen

Other

* No concurrent aspirin or other nonsteroidal anti-inflammatory drugs for ≥ 2 days before (5 days for drugs with a long half-life [e.g., naproxen, piraoxicam, difunisal, nabumetone, rofecoxib, or celecoxib] or 8 days for long acting agents), during, and for 2 days after completion of each pemetrexed disodium administration
* No concurrent participation in another study involving chemotherapy or radiotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-06-08 (Actual); Primary Completion 2011-04-29 (Actual); Study Completion 2017-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace K. Dy, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neoadjuvant Chemotherapy
Started | 38
Completed | 37
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Pathologically Complete Response
Description: Pathologic Complete Response is defined by a surgical pathology specimen, which is free of all gross and microscopic evidence of viable tumor.
Time Frame: 1 year
Population: ll treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 38
percentage of participants | 0 [0 to 9.2]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Frequency of Adverse Events, Graded According to NCI CTCAE v3.0. Please refer to the adverse event reporting for more detail.
Time Frame: 1 year
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 38
Participants
  Grade 1 | 2
  Grade 2 | 13
  Grade 3 | 19
  Grade 4 | 4

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as time from date of treatment initiation until date of death due to any cause.
Time Frame: Every 6 months until the time of death up to 126 months
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 38
months | 100.7 [37 to 126]

4. Secondary Outcome: Disease Free Survival
Description: Progressive disease is defined as at least a 20% increase in the sum of the longest diameter of target lesions or the appearance of new lesions. Disease Free Survival was defined as time from date of treatment initiation until date of first documented progression or date of death from any cause, whichever came first.
Time Frame: At least every 3 months after the completion of adjuvant therapy for two years and thereafter every 6 months for 3 years and then yearly up to 126 months
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 38
months | 34.5 [14.7 to 126]

5. Secondary Outcome: Correlation Between Response and Markers Such as Presence or Absence of ERCC1 and DHFR, TS, DPD and GARFT
Time Frame: 1 year
Population: No participants were analyzed as there was no budget left to do the analysis.
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 0

6. Secondary Outcome: Percent Change in SUV Level Between Pre and Post Chemotherapy
Description: Percent change of PET/SUV levels between baseline and post-chemotherapy.
Time Frame: Baseline and post-chemotherapy
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Percentage change in SUV level
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 38
Percentage change in SUV level | -36.1 (40.6)

ADVERSE EVENTS:
Arm/Group | Neoadjuvant Chemotherapy
Serious Adverse Events (participants affected / at risk) | 14/38
Other Adverse Events (participants affected / at risk) | 37/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Chemotherapy (N=38)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Empyema (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1)
Arterial thrombosis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Chemotherapy (N=38)
Anaemia (Blood and lymphatic system disorders) | 19 (22)
Leukopenia (Blood and lymphatic system disorders) | 12 (18)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 10 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (7)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2)
Ear congestion (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 10 (11)
Dry eye (Eye disorders) | 1 (1)
Eye discharge (Eye disorders) | 1 (1)
Eye irritation (Eye disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 12 (15)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Ileus paralytic (Gastrointestinal disorders) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 23 (33)
Reflux gastritis (Gastrointestinal disorders) | 1 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 4 (5)
Vomiting (Gastrointestinal disorders) | 8 (8)
Asthenia (General disorders) | 3 (3)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 3 (3)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 25 (35)
Feeling jittery (General disorders) | 1 (1)
Influenza like illness (General disorders) | 3 (3)
Injection site swelling (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 4 (4)
Pain (General disorders) | 3 (4)
Pyrexia (General disorders) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 5 (5)
Sinusitis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (4)
Blood alkaline phosphatase increased (Investigations) | 5 (5)
Haemoglobin (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 20 (41)
Hyperkalaemia (Metabolism and nutrition disorders) | 9 (12)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (4)
Dysgeusia (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 4 (5)
Hypoaesthesia (Nervous system disorders) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Vocal cord paresis (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5)
Panic attack (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (13)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sinusitis noninfective (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes